CLINICAL TRIAL: NCT05019131
Title: Addressing Provider Stress and Unconscious Bias to Improve Quality of Maternal Health Care
Brief Title: Caring for Providers to Improve Patient Experience Study Phase 2 in Migori County
Acronym: CPIPE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Kenya Medical Research Institute (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: A135552; R00HD093798 (NIH)
Record Dates: First submitted 2021-08-18; First posted 2021-08-24 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Maternal Health; Mental Health; Healthcare Provider; Adverse Outcomes; Stress; Stress, Psychological; Stress, Emotional; Quality of Care; Burnout; Discrimination, Social
Keywords: providers; mental health; unconscious bias; prejudice; Kenya; stress; burnout; person-centered care; quality of care; discrimination
MeSH Terms: conditions — Psychological Well-Being; Stress, Psychological; Burnout, Psychological; Social Discrimination; Bias, Implicit; Prejudice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): 1. Training: The investigators will develop a training for providers that addresses the following topics: Stress & positive coping mechanisms; Unconscious bias awareness and mitigation; Person-centered maternity care; Dealing with difficult situations; and Teamwork and communication;
  2. Peer support and mentorship: The investigators will identify what works best for these groups in terms of group composition, size, and how the groups want to interact.
  3. Leadership engagement: To ensure leadership buy in, support and sustainability of the intervention, the investigators will engage leadership of the County.
  4. Embedded champions: To facilitate ongoing engagement, the investigators will identify local leaders, and invite them to training where they will be taught how to facilitate peer support groups and serve as champions.
  Interventions: Behavioral: Training; Behavioral: Peer support and mentorship; Behavioral: Leadership engagement; Behavioral: Embedded champions
- Control arm (No Intervention): Will not receive any training during the intervention period

INTERVENTIONS:
Behavioral: Training — trainings to reduce conscious bias and stress
  Arms: Intervention arm
Behavioral: Peer support and mentorship — facilitated peer and mentorship opportunities
  Arms: Intervention arm
Behavioral: Leadership engagement — Engaged leadership at the county and facility levels
  Arms: Intervention arm
Behavioral: Embedded champions — Facilitate local champions to promote intervention
  Arms: Intervention arm

SUMMARY:
The activities described in this proposal are aimed at addressing health care provider stress and unconscious bias to improve quality of maternal health care, particularly related to the person-centered dimensions of care-i.e. care that is respectful and responsive to women's needs, preferences, and values. The investigators focus on health provider stress and unconscious bias because they are key drivers of poor-quality care that are often not addressed in interventions designed to improve quality of maternal health care. The investigators plan to (1) design an intervention that enables providers to identify and manage their stress and unconscious bias; (2) pilot the intervention to assess its feasibility and acceptability; and (3) assess preliminary effect of the intervention on: (a) provider knowledge, attitudes, and behaviors related to stress and unconscious bias; and (b) provider stress levels.

DETAILED DESCRIPTION:
Poor person-centered maternal health care (PCMHC) contributes to high maternal and neonatal mortality in sub-Saharan Africa (SSA), and disparities in PCMHC are driving disparities in use of maternal health services., However, little research exists on how to improve PCMHC and reduce disparities. The investigators seek to fill this gap with this project. They propose targeting health provider stress and unconscious bias as fundamental factors driving both poor PCMHC and disparities in PCMHC. Health care provider stress and unconscious bias are important to consider because: (1) providers in low-resource settings often work under very stressful conditions; (2) unconscious bias is prevalent in every society including SSA; and (3) these factors are mutually reinforcing drivers of poor quality care and disparities in person-centered care. In the first phase of the project (CPIPE1), they conducted research to examine (1) the factors associated with PCMHC and identified provider stress and unconscious bias as key contributing factors. They also examined the levels of provider stress and unconscious bias and the types of stressors and biases in Migori County, Kenya. The results of that research will be used to inform this phase (CPIPE2), the aims of which are to: (1) design a multicomponent theory and evidence-based intervention that enables providers to identify and manage their stress and unconscious bias; (2) pilot the intervention to assess its feasibility and acceptability; and (3) assess preliminary effect of the intervention on: (a) provider knowledge, attitudes, and behaviors related to stress and unconscious bias; and (b) provider stress levels using a pretest-posttest control group design. They will use the results of the pilot to refine the intervention and develop an R01 proposal for a multi-site evaluation with a larger sample and longer follow up to assess impact on PCMHC. This study will yield valuable information to inform quality improvement efforts for PCMHC.

ELIGIBILITY:
Inclusion Criteria:

* Providers working in maternity units of the intervention facilities are all eligible.

Exclusion Criteria:

* Inability to attend scheduled training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patience Afulani, PhD, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Migori County hospital and sub-county hospitals, Migori, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] WHO, UNICEF, UNFPA, The World Bank, United Nations Population Division. Trends in maternal mortality: 1990 to 2013 [Internet]. WHO. 2014 [cited 2014 Jul 17]. Available from: http://www.who.int/reproductivehealth/publications/monitoring/9789241503631/en/index.html
- [Background] Gabrysch S, Campbell OM. Still too far to walk: literature review of the determinants of delivery service use. BMC Pregnancy Childbirth. 2009 Aug 11;9:34. doi: 10.1186/1471-2393-9-34. PMID 19671156
- [Background] Moyer CA, Mustafa A. Drivers and deterrents of facility delivery in sub-Saharan Africa: a systematic review. Reprod Health. 2013 Aug 20;10:40. doi: 10.1186/1742-4755-10-40. PMID 23962135
- [Background] Graham WJ, McCaw-Binns A, Munjanja S. Translating coverage gains into health gains for all women and children: the quality care opportunity. PLoS Med. 2013;10(1):e1001368. doi: 10.1371/journal.pmed.1001368. Epub 2013 Jan 15. PMID 23335862
- [Background] van den Broek NR, Graham WJ. Quality of care for maternal and newborn health: the neglected agenda. BJOG. 2009 Oct;116(Suppl 1):18-21. doi: 10.1111/j.1471-0528.2009.02333.x. PMID 19740165
- [Background] Bohren MA, Hunter EC, Munthe-Kaas HM, Souza JP, Vogel JP, Gulmezoglu AM. Facilitators and barriers to facility-based delivery in low- and middle-income countries: a qualitative evidence synthesis. Reprod Health. 2014 Sep 19;11(1):71. doi: 10.1186/1742-4755-11-71. PMID 25238684
- [Background] Friberg IK, Kinney MV, Lawn JE, Kerber KJ, Odubanjo MO, Bergh AM, Walker N, Weissman E, Chopra M, Black RE; Science in Action: Saving the lives of Africa's Mothers, Newborns, and Children working group; Axelson H, Cohen B, Coovadia H, Diab R, Nkrumah F. Sub-Saharan Africa's mothers, newborns, and children: how many lives could be saved with targeted health interventions? PLoS Med. 2010 Jun 21;7(6):e1000295. doi: 10.1371/journal.pmed.1000295. PMID 20574515
- [Background] Miller S, Abalos E, Chamillard M, Ciapponi A, Colaci D, Comande D, Diaz V, Geller S, Hanson C, Langer A, Manuelli V, Millar K, Morhason-Bello I, Castro CP, Pileggi VN, Robinson N, Skaer M, Souza JP, Vogel JP, Althabe F. Beyond too little, too late and too much, too soon: a pathway towards evidence-based, respectful maternity care worldwide. Lancet. 2016 Oct 29;388(10056):2176-2192. doi: 10.1016/S0140-6736(16)31472-6. Epub 2016 Sep 16. PMID 27642019
- [Background] Leavitt M. Medscape's response to the Institute of Medicine Report: Crossing the quality chasm: a new health system for the 21st century. MedGenMed. 2001 Mar 5;3(2):2. No abstract available. PMID 11549951
- [Background] Bohren MA, Vogel JP, Hunter EC, Lutsiv O, Makh SK, Souza JP, Aguiar C, Saraiva Coneglian F, Diniz AL, Tuncalp O, Javadi D, Oladapo OT, Khosla R, Hindin MJ, Gulmezoglu AM. The Mistreatment of Women during Childbirth in Health Facilities Globally: A Mixed-Methods Systematic Review. PLoS Med. 2015 Jun 30;12(6):e1001847; discussion e1001847. doi: 10.1371/journal.pmed.1001847. eCollection 2015 Jun. PMID 26126110
- [Background] Abuya T, Warren CE, Miller N, Njuki R, Ndwiga C, Maranga A, Mbehero F, Njeru A, Bellows B. Exploring the prevalence of disrespect and abuse during childbirth in Kenya. PLoS One. 2015 Apr 17;10(4):e0123606. doi: 10.1371/journal.pone.0123606. eCollection 2015. PMID 25884566
- [Background] Moyer CA, Adongo PB, Aborigo RA, Hodgson A, Engmann CM. 'They treat you like you are not a human being': maltreatment during labour and delivery in rural northern Ghana. Midwifery. 2014 Feb;30(2):262-8. doi: 10.1016/j.midw.2013.05.006. Epub 2013 Jun 19. PMID 23790959
- [Background] Tuncalp O, Hindin MJ, Adu-Bonsaffoh K, Adanu R. Listening to women's voices: the quality of care of women experiencing severe maternal morbidity, in Accra, Ghana. PLoS One. 2012;7(8):e44536. doi: 10.1371/journal.pone.0044536. Epub 2012 Aug 31. PMID 22952992
- [Background] Koblinsky M, Moyer CA, Calvert C, Campbell J, Campbell OM, Feigl AB, Graham WJ, Hatt L, Hodgins S, Matthews Z, McDougall L, Moran AC, Nandakumar AK, Langer A. Quality maternity care for every woman, everywhere: a call to action. Lancet. 2016 Nov 5;388(10057):2307-2320. doi: 10.1016/S0140-6736(16)31333-2. Epub 2016 Sep 16. PMID 27642018
- [Background] Ratcliffe HL, Sando D, Lyatuu GW, Emil F, Mwanyika-Sando M, Chalamilla G, Langer A, McDonald KP. Mitigating disrespect and abuse during childbirth in Tanzania: an exploratory study of the effects of two facility-based interventions in a large public hospital. Reprod Health. 2016 Jul 18;13(1):79. doi: 10.1186/s12978-016-0187-z. PMID 27424608
- [Background] Ratcliffe HL, Sando D, Mwanyika-Sando M, Chalamilla G, Langer A, McDonald KP. Applying a participatory approach to the promotion of a culture of respect during childbirth. Reprod Health. 2016 Jul 18;13(1):80. doi: 10.1186/s12978-016-0186-0. PMID 27424514
- [Background] Filby A, McConville F, Portela A. What Prevents Quality Midwifery Care? A Systematic Mapping of Barriers in Low and Middle Income Countries from the Provider Perspective. PLoS One. 2016 May 2;11(5):e0153391. doi: 10.1371/journal.pone.0153391. eCollection 2016. PMID 27135248
- [Background] UNC Executive Development. The Real Effects of Unconscious Bias in the Workplace [Internet]. 2015 [cited 2016 Oct 26]. Available from: http://execdev.kenan-flagler.unc.edu/blog/the-real-effects-of-unconscious-bias-in-the-workplace-0
- [Background] Leape LL, Shore MF, Dienstag JL, Mayer RJ, Edgman-Levitan S, Meyer GS, Healy GB. Perspective: a culture of respect, part 1: the nature and causes of disrespectful behavior by physicians. Acad Med. 2012 Jul;87(7):845-52. doi: 10.1097/ACM.0b013e318258338d. PMID 22622217
- [Background] Leape LL, Shore MF, Dienstag JL, Mayer RJ, Edgman-Levitan S, Meyer GS, Healy GB. Perspective: a culture of respect, part 2: creating a culture of respect. Acad Med. 2012 Jul;87(7):853-8. doi: 10.1097/ACM.0b013e3182583536. PMID 22622219
- [Background] Andersen HM. "Villagers": differential treatment in a Ghanaian hospital. Soc Sci Med. 2004 Nov;59(10):2003-12. doi: 10.1016/j.socscimed.2004.03.005. PMID 15351468
- [Background] Glanz K, Rimer KB. Theory at a Glance: A Guide for Health Promotion Practice. National Cancer Institute, National Institutes of Health, U.S. Department of Health and Human Services. NIH Pub. No. 97-3896. Washington, DC: NIH. 1997.
- [Background] San Francisco Department of Public Health. Trauma Informed Systems Initiative 2014 Year in Review [Internet]. 2015. Available from: http://www.leapsf.org/pdf/Trauma-Informed-Systems-Initative-2014.pdf
- [Background] McLeroy KR, Bibeau D, Steckler A, Glanz K. An ecological perspective on health promotion programs. Health Educ Q. 1988 Winter;15(4):351-77. doi: 10.1177/109019818801500401. PMID 3068205
- [Background] Alkema L, Chou D, Hogan D, Zhang S, Moller AB, Gemmill A, Fat DM, Boerma T, Temmerman M, Mathers C, Say L; United Nations Maternal Mortality Estimation Inter-Agency Group collaborators and technical advisory group. Global, regional, and national levels and trends in maternal mortality between 1990 and 2015, with scenario-based projections to 2030: a systematic analysis by the UN Maternal Mortality Estimation Inter-Agency Group. Lancet. 2016 Jan 30;387(10017):462-74. doi: 10.1016/S0140-6736(15)00838-7. Epub 2015 Nov 13. PMID 26584737
- [Background] WHO. PMNCH Fact Sheet: Maternal mortality [Internet]. 2011 [cited 2013 Jul 16]. Available from: http://www.who.int/pmnch/media/press_materials/fs/fs_mdg5_maternalmortality/en/index.html
- [Background] WHO. Making pregnancy safer: the critical role of the skilled attendant. Jt Statement WHO ICM FIGO Geneva. 2004;
- [Background] Khan KS, Wojdyla D, Say L, Gulmezoglu AM, Van Look PF. WHO analysis of causes of maternal death: a systematic review. Lancet. 2006 Apr 1;367(9516):1066-1074. doi: 10.1016/S0140-6736(06)68397-9. PMID 16581405
- [Background] Say L, Chou D, Gemmill A, Tuncalp O, Moller AB, Daniels J, Gulmezoglu AM, Temmerman M, Alkema L. Global causes of maternal death: a WHO systematic analysis. Lancet Glob Health. 2014 Jun;2(6):e323-33. doi: 10.1016/S2214-109X(14)70227-X. Epub 2014 May 5. PMID 25103301
- [Background] WHO. Global Health Observatory Data Repository, MDG 5: Maternal health: [Internet]. 2013 [cited 2013 Sep 5]. Available from: http://apps.who.int/gho/data/node.main.REPWOMEN39
- [Background] March of Dimes, PMNCH, Save the Children. Born Too Soon: The Global Action Report on Preterm Birth. Eds CP Howson, MV Kinney, JE Lawn. World Health Organization, Geneva; 2012.
- [Background] Kenya National Bureau of Statistics, Ministry of Health, National AIDS Control Council, Kenya Medical Research Institute, National Council for Population and Development, Nairobi, Kenya, and The DHS Program, ICF International, Rockville, Maryland, USA. The DHS Program - Kenya: DHS, 2014 - Final Report (English) [Internet]. 2015 [cited 2016 Feb 18]. Available from: http://dhsprogram.com/publications/publication-FR308-DHS-Final-Reports.cfm
- [Background] Anwar I, Kalim N, Koblinsky M. Quality of obstetric care in public-sector facilities and constraints to implementing emergency obstetric care services: evidence from high- and low-performing districts of Bangladesh. J Health Popul Nutr. 2009 Apr;27(2):139-55. doi: 10.3329/jhpn.v27i2.3327. PMID 19489412
- [Background] Afulani PA, Kirumbi L, Lyndon A. What makes or mars the facility-based childbirth experience: thematic analysis of women's childbirth experiences in western Kenya. Reprod Health. 2017 Dec 29;14(1):180. doi: 10.1186/s12978-017-0446-7. PMID 29284490
- [Background] Afulani PA, Moyer C. Explaining Disparities in Use of Skilled Birth Attendants in Developing Countries: A Conceptual Framework. PLoS One. 2016 Apr 22;11(4):e0154110. doi: 10.1371/journal.pone.0154110. eCollection 2016. PMID 27105309
- [Background] Fahy K. What is woman-centred care and why does it matter? Women Birth. 2012 Dec;25(4):149-51. doi: 10.1016/j.wombi.2012.10.005. No abstract available. PMID 23177665
- [Background] Pope R, Graham L, Patel S. Woman-centred care. Int J Nurs Stud. 2001 Apr;38(2):227-38. doi: 10.1016/s0020-7489(00)00034-1. PMID 11223063
- [Background] Downe S, Lawrie TA, Finlayson K, Oladapo OT. Effectiveness of respectful care policies for women using routine intrapartum services: a systematic review. Reprod Health. 2018 Feb 6;15(1):23. doi: 10.1186/s12978-018-0466-y. PMID 29409519
- [Background] Rubashkin N, Warnock R, Diamond-Smith N. A systematic review of person-centered care interventions to improve quality of facility-based delivery. Reprod Health. 2018 Oct 10;15(1):169. doi: 10.1186/s12978-018-0588-2. PMID 30305129
- [Background] Abuya T, Ndwiga C, Ritter J, Kanya L, Bellows B, Binkin N, Warren CE. The effect of a multi-component intervention on disrespect and abuse during childbirth in Kenya. BMC Pregnancy Childbirth. 2015 Sep 22;15:224. doi: 10.1186/s12884-015-0645-6. PMID 26394616
- [Background] Familoni OB. An overview of stress in medical practice. Afr Health Sci. 2008 Mar;8(1):6-7. No abstract available. PMID 19357725
- [Background] Yeboah MA, Ansong MO, Antwi HA, Yiranbon E, Anyan F, Gyebil F. Determinants of Workplace Stress among Healthcare Professionals in Ghana: An Empirical Analysis. ResearchGate. 2014 Mar 1;Vol. 5(No. 4 [Special Issue]):140-151.
- [Background] Cooper LA, Roter DL, Carson KA, Beach MC, Sabin JA, Greenwald AG, Inui TS. The associations of clinicians' implicit attitudes about race with medical visit communication and patient ratings of interpersonal care. Am J Public Health. 2012 May;102(5):979-87. doi: 10.2105/AJPH.2011.300558. Epub 2012 Mar 15. PMID 22420787
- [Background] Nosek BA, Ranganath KA, Smith CT, Chugh D, Olson KR, Lindner NM, Greenwald AG, Devos T, Banaji M, Smyth FL, Hansen JJ. Pervasiveness and Correlates of Implicit Attitudes and Stereotypes. 2007 [cited 2016 Dec 8]; Available from: https://dash.harvard.edu/handle/1/2958438
- [Background] Blair IV, Steiner JF, Havranek EP. Unconscious (implicit) bias and health disparities: where do we go from here? Perm J. 2011 Spring;15(2):71-8. doi: 10.7812/TPP/11.979. PMID 21841929
- [Background] Major B, Mendes WB, Dovidio JF. Intergroup relations and health disparities: a social psychological perspective. Health Psychol. 2013 May;32(5):514-24. doi: 10.1037/a0030358. PMID 23646834
- [Background] Chapman EN, Kaatz A, Carnes M. Physicians and implicit bias: how doctors may unwittingly perpetuate health care disparities. J Gen Intern Med. 2013 Nov;28(11):1504-10. doi: 10.1007/s11606-013-2441-1. Epub 2013 Apr 11. PMID 23576243
- [Background] McEwen BS. Stressed or stressed out: what is the difference? J Psychiatry Neurosci. 2005 Sep;30(5):315-8. PMID 16151535
- [Background] Public Health England. Interventions to prevent burnout in high risk individuals: evidence review - Publications - GOV.UK [Internet]. 2016 [cited 2016 Oct 26]. Available from: https://www.gov.uk/government/publications/interventions-to-prevent-burnout-in-high-risk-individuals-evidence-review
- [Background] Halbesleben JRB, editor. Handbook of Stress and Burnout in Health Care. 3 edition. New York: Nova Science Pub Inc; 2008.
- [Background] Wallace JE, Lemaire JB, Ghali WA. Physician wellness: a missing quality indicator. Lancet. 2009 Nov 14;374(9702):1714-21. doi: 10.1016/S0140-6736(09)61424-0. PMID 19914516
- [Background] Klein J, Grosse Frie K, Blum K, von dem Knesebeck O. Burnout and perceived quality of care among German clinicians in surgery. Int J Qual Health Care. 2010 Dec;22(6):525-30. doi: 10.1093/intqhc/mzq056. Epub 2010 Oct 8. PMID 20935011
- [Background] Krasner MS, Epstein RM, Beckman H, Suchman AL, Chapman B, Mooney CJ, Quill TE. Association of an educational program in mindful communication with burnout, empathy, and attitudes among primary care physicians. JAMA. 2009 Sep 23;302(12):1284-93. doi: 10.1001/jama.2009.1384. PMID 19773563
- [Background] Shanafelt TD, Sloan JA, Habermann TM. The well-being of physicians. Am J Med. 2003 Apr 15;114(6):513-9. doi: 10.1016/s0002-9343(03)00117-7. No abstract available. PMID 12727590
- [Background] Khalil D. Violence against midwives in Cape Town. Afr J Midwifery Womens Health. 2009 Feb 1;3(1):37-40.
- [Background] Fauveau V, Sherratt DR, de Bernis L. Human resources for maternal health: multi-purpose or specialists? Hum Resour Health. 2008 Sep 30;6:21. doi: 10.1186/1478-4491-6-21. PMID 18826600
- [Background] Afulani PA, Kelly AM, Buback L, Asunka J, Kirumbi L, Lyndon A. Providers' perceptions of disrespect and abuse during childbirth: a mixed-methods study in Kenya. Health Policy Plan. 2020 Jun 1;35(5):577-586. doi: 10.1093/heapol/czaa009. PMID 32154878
- [Background] Mendes WB, Koslov K. Brittle smiles: positive biases toward stigmatized and outgroup targets. J Exp Psychol Gen. 2013 Aug;142(3):923-33. doi: 10.1037/a0029663. Epub 2012 Aug 13. PMID 22889160
- [Background] Green AR, Carney DR, Pallin DJ, Ngo LH, Raymond KL, Iezzoni LI, Banaji MR. Implicit bias among physicians and its prediction of thrombolysis decisions for black and white patients. J Gen Intern Med. 2007 Sep;22(9):1231-8. doi: 10.1007/s11606-007-0258-5. Epub 2007 Jun 27. PMID 17594129
- [Background] Sabin JA, Greenwald AG. The influence of implicit bias on treatment recommendations for 4 common pediatric conditions: pain, urinary tract infection, attention deficit hyperactivity disorder, and asthma. Am J Public Health. 2012 May;102(5):988-95. doi: 10.2105/AJPH.2011.300621. Epub 2012 Mar 15. PMID 22420817
- [Background] Turan JM, Hatcher AH, Medema-Wijnveen J, Onono M, Miller S, Bukusi EA, Turan B, Cohen CR. The role of HIV-related stigma in utilization of skilled childbirth services in rural Kenya: a prospective mixed-methods study. PLoS Med. 2012;9(8):e1001295. doi: 10.1371/journal.pmed.1001295. Epub 2012 Aug 21. PMID 22927800
- [Background] Turan JM, Bukusi EA, Onono M, Holzemer WL, Miller S, Cohen CR. HIV/AIDS stigma and refusal of HIV testing among pregnant women in rural Kenya: results from the MAMAS Study. AIDS Behav. 2011 Aug;15(6):1111-20. doi: 10.1007/s10461-010-9798-5. PMID 20827573
- [Background] Tincher MM, Lebois LA, Barsalou LW. Mindful attention reduces linguistic intergroup bias. Mindfulness (N Y). 2016 Apr;7(2):349-360. doi: 10.1007/s12671-015-0450-3. Epub 2015 Oct 15. PMID 27200110
- [Background] Devine PG, Forscher PS, Austin AJ, Cox WT. Long-term reduction in implicit race bias: A prejudice habit-breaking intervention. J Exp Soc Psychol. 2012 Nov;48(6):1267-1278. doi: 10.1016/j.jesp.2012.06.003. PMID 23524616
- [Background] Clarke AE. Situational Analysis: Grounded Theory After the Postmodern Turn. 1 edition. Thousand Oaks, Calif: SAGE Publications, Inc; 2005.
- [Background] Lateef F. Simulation-based learning: Just like the real thing. J Emerg Trauma Shock. 2010 Oct;3(4):348-52. doi: 10.4103/0974-2700.70743. PMID 21063557
- [Background] Sally S. Russell. An Overview of Adult Learning Processes [Internet]. Medscape. [cited 2016 Nov 7]. Available from: http://www.medscape.com/viewarticle/547417
- [Background] Bloom SL. Organizational Stress and Trauma-Informed Services. In: Levin BL, Becker MA, editors. Public Health Perspect Womens Ment Health [Internet]. Springer New York; 2010 [cited 2016 Dec 6]. p. 295-311. Available from: http://link.springer.com/chapter/10.1007/978-1-4419-1526-9_15
- [Background] Proctor EK, Powell BJ, Baumann AA, Hamilton AM, Santens RL. Writing implementation research grant proposals: ten key ingredients. Implement Sci. 2012 Oct 12;7:96. doi: 10.1186/1748-5908-7-96. PMID 23062065
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Carroll C, Patterson M, Wood S, Booth A, Rick J, Balain S. A conceptual framework for implementation fidelity. Implement Sci. 2007 Nov 30;2:40. doi: 10.1186/1748-5908-2-40. PMID 18053122
- [Background] Breitenstein SM, Gross D, Garvey CA, Hill C, Fogg L, Resnick B. Implementation fidelity in community-based interventions. Res Nurs Health. 2010 Apr;33(2):164-73. doi: 10.1002/nur.20373. PMID 20198637
- [Background] Rossi PH, Lipsey MW, Freeman HE. Evaluation: A systematic approach. 7th ed. Thousand Oaks, CA: Sage Publications, Inc.; 2004:68-81.
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Gerber M, Colledge F, Mucke M, Schilling R, Brand S, Ludyga S. Psychometric properties of the Shirom-Melamed Burnout Measure (SMBM) among adolescents: results from three cross-sectional studies. BMC Psychiatry. 2018 Aug 25;18(1):266. doi: 10.1186/s12888-018-1841-5. PMID 30144799
- [Background] Kim HG, Cheon EJ, Bai DS, Lee YH, Koo BH. Stress and Heart Rate Variability: A Meta-Analysis and Review of the Literature. Psychiatry Investig. 2018 Mar;15(3):235-245. doi: 10.30773/pi.2017.08.17. Epub 2018 Feb 28. PMID 29486547
- [Background] Jarvelin-Pasanen S, Sinikallio S, Tarvainen MP. Heart rate variability and occupational stress-systematic review. Ind Health. 2018 Nov 21;56(6):500-511. doi: 10.2486/indhealth.2017-0190. Epub 2018 Jun 16. PMID 29910218
- [Background] Lennartsson AK, Jonsdottir I, Sjors A. Low heart rate variability in patients with clinical burnout. Int J Psychophysiol. 2016 Dec;110:171-178. doi: 10.1016/j.ijpsycho.2016.08.005. Epub 2016 Aug 14. PMID 27535344
- [Background] Russell E, Koren G, Rieder M, Van Uum S. Hair cortisol as a biological marker of chronic stress: current status, future directions and unanswered questions. Psychoneuroendocrinology. 2012 May;37(5):589-601. doi: 10.1016/j.psyneuen.2011.09.009. Epub 2011 Oct 4. PMID 21974976
- [Background] Sauve B, Koren G, Walsh G, Tokmakejian S, Van Uum SH. Measurement of cortisol in human hair as a biomarker of systemic exposure. Clin Invest Med. 2007;30(5):E183-91. doi: 10.25011/cim.v30i5.2894. PMID 17892760
- [Background] Afulani PA, Diamond-Smith N, Golub G, Sudhinaraset M. Development of a tool to measure person-centered maternity care in developing settings: validation in a rural and urban Kenyan population. Reprod Health. 2017 Sep 22;14(1):118. doi: 10.1186/s12978-017-0381-7. PMID 28938885
- [Background] Afulani PA, Buback L, Kelly AM, Kirumbi L, Cohen CR, Lyndon A. Providers' perceptions of communication and women's autonomy during childbirth: a mixed methods study in Kenya. Reprod Health. 2020 Jun 3;17(1):85. doi: 10.1186/s12978-020-0909-0. PMID 32493424
- [Background] Lane, K. A., Banaji, M. R., Nosek, B. A. & Greenwald, A. G. Understanding and Using the Implicit Association Test: IV: What We Know (So Far) about the Method. in Implicit measures of attitudes (eds. Wittenbrink, B. & Schwarz, N.) 59-102 (Guilford Press, 2007).
- [Background] About the IAT. Available at: https://implicit.harvard.edu/implicit/iatdetails.html.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Health facilities participating in the study
Groups:
- Intervention Arm: 1. Training: The investigators will develop a training for providers that addresses the following topics: Stress & positive coping mechanisms; Unconscious bias awareness and mitigation; Person-centered maternity care; Dealing with difficult situations; and Teamwork and communication;
  2. Peer support and mentorship: The investigators will identify what works best for these groups in terms of group composition, size, and how the groups want to interact.
  3. Leadership engagement: To ensure leadership buy in, support and sustainability of the intervention, the investigators will engage leadership of the County.
  4. Embedded champions: To facilitate ongoing engagement, the investigators will identify local leaders, and invite them to training where they will be taught how to facilitate peer support groups and serve as champions.
  Training: trainings to reduce conscious bias and stress
  Peer support and mentorship: facilitated peer and mentorship opportunities
  Leadership engagement: Engaged leadership at the county and facility levels
  Embedded champions: Facilitate local champions to promote intervention
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 40 | 43
Completed | 40 | 40
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 40 | 43 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 43 | 83
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 29 | 61
  Male | 8 | 14 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 40 | 43 | 83
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Kenya | 40 | 43 | 83

OUTCOME MEASURES:

1. Primary Outcome: Change in Perceived Stress Scale (PSS) Score From Baseline to 6 Months
Description: The Perceived Stress Scale (PSS) score ranges from 0 to 40 with higher scores indicating higher perceived stress.
Time Frame: Baseline and 6 months
Population: health care providers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 40 | 40
score on a scale
  Baseline | 20.89 (3.86) | 20.58 (4.51)
  End line | 18.63 (5.34) | 20.05 (5.57)

2. Primary Outcome: Change in Shirom-Melamed Burnout Measure (SMBM) Score From Baseline to 6 Months
Description: The Shirom-Melamed Burnout Measure range from 1 to 7 with higher scores indicating higher burnout
Time Frame: Baseline and 6 months
Population: health care providers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 40 | 40
score on a scale
  Baseline | 3.64 (1.05) | 3.70 (1.10)
  End line | 2.95 (0.97) | 3.42 (1.08)

3. Primary Outcome: Change in Stress Knowledge and Attitudes Score From Baseline to 6 Months
Description: The stress knowledge and attitudes score is measured by 14 survey questions with scores ranging from 0 to 14. Higher scores indicate higher knowledge and positive attitudes regarding stress and stress management. We used 13 of the items from the 14-item survey scale. The score range used is 0 to 13- as noted in the limitations section.
Time Frame: Baseline and 6 months
Population: health care providers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 40 | 40
score on a scale
  Baseline | 7.78 (2.41) | 7.95 (2.77)
  End line | 9.50 (1.80) | 8.53 (2.01)

4. Primary Outcome: Change in Unconscious Bias Knowledge and Attitudes Score From Baseline to 6 Months
Description: The unconscious bias knowledge and attitudes score is measured by 17 survey questions with scores ranging from 0 to 17. Higher scores indicate higher knowledge and positive attitudes regarding unconscious bias and unconscious bias mitigation
Time Frame: Baseline and 6 months
Population: health care providers
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 40 | 40
score on a scale
  Baseline | 8.93 (1.94) | 9.13 (2.14)
  End line | 10.70 (1.73) | 9.45 (2.16)

5. Secondary Outcome: Change in Hair Cortisol Levels From Baseline to 6 Months
Description: There are no specified cut-offs for cortisol levels, but, on average, higher cortisol levels indicate higher stress.
Time Frame: Baseline and 6 months
Population: health care providers
Measure: Mean (Standard Deviation); unit: pg/mg
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 15 | 7
pg/mg
  Baseline | 74.13 (147.38) | 8.43 (3.03)
  End line | 41.50 (72.19) | 36.05 (58.29)

6. Secondary Outcome: Change in Heart Rate Variability (HRV) Levels From Baseline to 6 Months
Description: There are no specified cut-offs for HRV but, on average, lower HRV scores indicate higher stress
Time Frame: Baseline and 6 months
Population: health care providers
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 34 | 32
ms
  Baseline | 3.70 (0.59) | 3.71 (0.61)
  End line | 3.71 (0.43) | 3.84 (0.63)

7. Secondary Outcome: Change in Socioeconomic Status-person Centered Maternity Care Implicit Association Test (IAT) Score
Description: IAT scores vary between -2 and +2. For this study, higher positive scores indicates a stronger implicit association between high status with good patient and low status with difficult patient
Time Frame: Baseline and 6 months
Population: health care providers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 34 | 34
score on a scale
  Baseline | 0.75 (0.37) | 0.67 (0.46)
  End line | 0.62 (0.52) | 0.43 (0.55)

8. Secondary Outcome: Change in Explicit Bias Scores From Baseline to 6 Months
Description: The explicit bias scores are from responses to a vignette and range from 4 to 28. Higher scores indicate more explicit bias
Time Frame: Baseline and 6 months
Population: Health care providers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 40 | 40
score on a scale
  Baseline | 17.38 (3.06) | 16.30 (3.27)
  End line | 15.65 (3.76) | 14.91 (3.12)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/43
Other Adverse Events (participants affected / at risk) | 0/40 | 0/43

LIMITATIONS AND CAVEATS:
Our initial plan was to use 14 and 17 items for assessing stress and bias knowledge and attitudes respectively, but the final analysis used 13 and 15 items- 3 questions did not perform well during pretesting. Change in Hair Cortisol Levels includes for analysis the total number of participants we were able to collect hair samples with- 15 and 7, for intervention and control, respecively. Change in Heart Rate Variability (HRV) Levels were limited to those who consented and provided HRV data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/31/NCT05019131/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/31/NCT05019131/ICF_001.pdf